CLINICAL TRIAL: NCT05798182
Title: Ultrasound in the Intensive Care Unit and Measurable Indicators of Systemic Inflammation
Brief Title: Ultrasound Markers of Systemic Inflammation
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Sponsor
Other Study IDs: 2158-61-07-21-96
Record Dates: First submitted 2022-06-02; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2021-05

CONDITIONS: Inflammation Process; Endothelial Dysfunction; Vasomotor Arterial Disorder; Vascular Dilation; Swelling; Hand
Keywords: Intensive Care, Surgical; Ultrasonography, Doppler; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients: Adult patients admitted to the ICU.
  Interventions: Diagnostic Test: Ultrasound measurement

INTERVENTIONS:
Diagnostic Test: Ultrasound measurement — Study was conducted with Mindray T7 ultrasound machine using linear probe. Vascular ultrasound mode was used with settings depth of 50 mm and gain of 40 dB during the entire study period. The diameter and flow velocity of the brachial artery and wrist edema of the fist were measured within 24 hours of admission and the following day.
  Other Names: Mindray T7 ultrasound machine

SUMMARY:
The aim of this study was to measure whether the flow rate through the brachial artery and inflammatory markers were associated with the development of tissue edema in the surgical intensive care unit patients.

DETAILED DESCRIPTION:
The study was performed using a ultrasound machine with linear probe settings at 50 mm depth and 40 decibel [dB] gain that did not change during the study. The probe was placed on vascular ultrasound measurement. The diameter of the brachial artery in the middle of the upper arm and the flow rate through the artery was measured on postoperative days 1 and 2. The presence of the edema was measured above the 3rd metacarpal bone as the distance from the skin surface to the periosteum. An average of three assessments was shown. Patient's age, body mass index (BMI), type of admission, white blood cells (WBC), C-reactive protein (CRP), and procalcitonin (PCT) were also registered.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Postoperative surgical patients
* Signed informed consent

Exclusion Criteria:

* Refusal to give informed consent
* A previous thromboembolic event of the brachial artery
* Acute infection of the upper extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in Osijek University Hospital who are admitted in the ICU will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Diameter of brachial artery - 1 | within 4 hours of admission.
  Measurement of a brachial artery diameter [cm] at admission. Admission day is considered as day 1.
Diameter of brachial artery - 2 | day 2 after admission is between 24 and 48 hours after admission.
  measurement of a brachial artery diameter [cm] on day 2 after admission.
Brachial artery flow velocity - 1 | within 4 hours of admission to ICU.
  measurement of a brachial artery flow velocity [cm/s] at admission.
Brachial artery flow velocity - 2 | day 2 after admission is between 24 and 48 hours after admission.
  measurement of a brachial artery flow velocity [cm/s] on day 2 after admission. Day 2 is Measurement of a brachial artery flow velocity [cm/s] between 24 and 48 h after ICU admission.
Distance from skin to third metacarpal bone -1 | within 4 hours of admission.
  measurement of a distance from the skin to third metacarpal bone (cm) at admission.
Distance from skin to third metacarpal bone - 2 | day 2 after admission is between 24 and 48 hours after admission.
  measurement of a distance from the skin to third metacarpal bone (cm) on day 2 after admission.
White blood cell count - 1 | within 4 hours of admission.
  blood sample analysis for white blood cell count (WBC [10^9/L]) at admission.
White blood cell count - 2 | day 2 after admission is between 24 and 48 hours after admission.
  blood sample analysis for white blood cell count (WBC [10^9/L]) on day 2 after admission.
C-reactive protein - 1 | within 4 hours of admission.
  blood sample analysis for C-reactive protein (CRP [mg/L]) concentration at admission.
C-reactive protein - 2 | day 2 after admission is between 24 and 48 hours after admission.
  Blood sample analysis for C-reactive protein (CRP [mg/L]) concentration on day 2 after admission.
Procalcitonin - 1 | within 4 hours of admission.
  blood sample analysis for Procalcitonin concentration (PCT [ug/L]) at admission.
Procalcitonin - 2 | Day 2 after admission is between 24 and 48 hours after admission.
  Blood sample analysis for Procalcitonin concentration (PCT [ug/L]) on day 2 after admission.

CONTACTS AND LOCATIONS:
Overall Officials: Slavica Kvolik, M.D., PhD,, Study Director — Osijek University Hospital
Locations (1):
- Slavica Kvolik, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chakraborty RK, Burns B. Systemic Inflammatory Response Syndrome. [Updated 2021 Jul 28]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2022 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK547669/
- [Background] Čavka A, Tadžić R, Grizelj I, Unfirer S, Mihaljević Z, Mihalj M et al. Endotelna funkcija - funkcionalni pokazatelj kardiovaskularnih rizičnih čimbenika. Medicinski vjesnik [Internet]. 2012 [Accessed 23.05.2021.];44((1-4)):135-146. Available from: https://hrcak.srce.hr/187756
- [Background] Lu D, Kassab GS. Role of shear stress and stretch in vascular mechanobiology. J R Soc Interface. 2011 Oct 7;8(63):1379-85. doi: 10.1098/rsif.2011.0177. Epub 2011 Jul 6. PMID 21733876
- [Background] Chen L, Deng H, Cui H, Fang J, Zuo Z, Deng J, Li Y, Wang X, Zhao L. Inflammatory responses and inflammation-associated diseases in organs. Oncotarget. 2017 Dec 14;9(6):7204-7218. doi: 10.18632/oncotarget.23208. eCollection 2018 Jan 23. PMID 29467962
- [Background] Mortaz E, Alipoor SD, Adcock IM, Mumby S, Koenderman L. Update on Neutrophil Function in Severe Inflammation. Front Immunol. 2018 Oct 2;9:2171. doi: 10.3389/fimmu.2018.02171. eCollection 2018. PMID 30356867
- [Background] Sproston NR, Ashworth JJ. Role of C-Reactive Protein at Sites of Inflammation and Infection. Front Immunol. 2018 Apr 13;9:754. doi: 10.3389/fimmu.2018.00754. eCollection 2018. PMID 29706967
- [Background] Evans DH. Colour flow and motion imaging. Proc Inst Mech Eng H. 2010;224(2):241-53. doi: 10.1243/09544119JEIM599. PMID 20349817
- [Background] Kubler A, Maciejewski D, Adamik B, Kaczorowska M. Mechanical ventilation in ICUs in Poland: a multi-center point-prevalence study. Med Sci Monit. 2013 Jun 3;19:424-9. doi: 10.12659/MSM.883930. PMID 23727991